CLINICAL TRIAL: NCT02244723
Title: Prospective, Observational Study of Diagnostic Value of Lung Ultrasound for Ventilator-Associated Pneumonia
Brief Title: Diagnostic Value of Lung Ultrasound for Ventilator-Associated Pneumonia
Acronym: VPLUS
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Principal Investigator, bélaid BOUHEMAD, M.D., Fondation Hôpital Saint-Joseph
Other Study IDs: VPLUS
Record Dates: First submitted 2013-09-05; First posted 2014-09-19 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Ventilator-Associated Pneumonia; diagnosis
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Biochemical data (WBC count with differential, arterial blood gas)
  * Microbiological data (UTA and BAL) - UTA data must have been collected within 24 hours of enrollment and BAL data within 12 hours of enrollment (unprotected tracheal aspirate (UTA)- fibrobronchoscopy with protected distal sampling)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected VAP: Only one group is studied : mechanically-ventilated patients with suspected VAP in ICUs.
  For each patient a lung ultrasound examination will be performed.
  Interventions: Other: Lung ultrasound examination

INTERVENTIONS:
Other: Lung ultrasound examination — Lung ultrasound (LUS) is increasingly being used at the bedside for assessing alveolar-interstitial syndrome, lung consolidation, pneumonia, pneumothorax, and pleural effusion. It could be an easily repeatable noninvasive tool for diagnosis of ventilator associated pneumonia

SUMMARY:
Ventilator-associated pneumonia (VAP) is the most common nosocomial infection acquired by mechanically-ventilated patients in the intensive care unit (ICU). It has significant clinical and economic consequences, as it is associated with considerable morbidity, increased mortality, and excess health care costs. Appropriate antibiotic therapy for patients with VAP significantly improves outcomes, making rapid identification of patients with VAP an important clinical goal.

This application is for support of a prospective, multi-centered study to evaluate the diagnostic value of lung ultrasound for VAP. The primary hypothesis is that the association of the Clinical Pulmonary Infection Score (CPIS) to specific lung ultrasound signs could allow for early and reliable diagnosis of bacterial VAP.

Objective 1: To evaluate the sensitivity, specificity, and diagnostic accuracy of lung ultrasound alone and in association with the CPIS.

Objective 2: To determine the frequency of specific lung ultrasound signs (subpleural consolidation, irregular B-lines) in VAP.

Objective 3: To promote development of a diagnostic pathway for VAP incorporating CPIS, lung ultrasound, and unprotected tracheal aspirate (UTA).

DETAILED DESCRIPTION:
Patients will be enrolled within 24 hours of the point at which criteria are met for suspected VAP. Upon enrollment, the following variables will be recorded from the online medical record, and a Clinical Pulmonary Infection Score will be calculated.

* Demographics (height, weight, comorbidities)
* Ventilation parameters
* Infectious disease data during present admission (antibiotic history, culture data)
* Biochemical data (WBC count with differential, arterial blood gas)
* Microbiological data (UTA and BAL) - UTA data must have been collected within 24 hours of enrollment and BAL data within 12 hours of enrollment
* Radiological data (CXR or chest CT)

Lung ultrasound will be performed within 24 hours of the point at which criteria are met for suspected VAP. Lung ultrasound will include examination of both lungs. Each hemithorax will be divided into three regions using anterior and posterior axillary lines as landmarks. Each of these regions will be further divided into upper and lower quadrants, yielding a total of 6 quadrants per hemithorax. Examination will specifically identify the presence or absence of the following lung ultrasound findings: normal pleural A lines, non-coalescent B lines, coalescent B lines, consolidations (subpleural or lobar), and linear air bronchograms. A Lung Ultrasound Aeration Score will be calculated based on these findings. Ultrasonographic diagnosis of VAP will be defined based on the presence of subpleural consolidation, entire lobar consolidation, or air bronchogram within consolidation.

The results of microbiological data will be followed up for confirmation of culture results. Cultures will be considered positive if ≥ 100,000 bacterial colony-forming units (cfu) are isolated.

At day #28 of study enrollment, the patient's status will be documented (alive vs. deceased, inpatient vs. discharged).

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation for at least 48 hours,
* New or evolving infiltrate on chest radiograph (CXR) or computed tomography (CT), and
* A minimum of two of the following clinical criteria:

  * Body temperature ≥ 38.5° C (101° F) or < 36° C (97° F)
  * White blood cell count > 10,000/ml or < 4,000/ml or > 10% immature cells
  * Partial pressure of oxygen in arterial blood < 60 mmHg or partial pressure of oxygen in arterial blood/ inspired oxygen fraction ratio < 300
  * Purulent respiratory secretions

Exclusion Criteria:

Known ongoing pneumonia

* Patient younger than 18 years old
* Mechanical ventilation <48 hours
* Contraindication to bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects will be recruited from mechanically-ventilated patients with suspected VAP in ICUs
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
ventilator-associated pneumonia. | up to 30days
  Ventilator associated pneumonia is diagnosed when patient has a positive broncho alveolar lavage (positive cultiure >10*3 CFU/ml) and clinical criteria (◦Body temperature ≥ 38.5° C (101° F) or < 36° C (97° F)
  * White blood cell count > 10,000/ml or < 4,000/ml or > 10% immature cells
  * Partial pressure of oxygen in arterial blood < 60 mmHg or partial pressure of oxygen in arterial blood/ inspired oxygen fraction ratio < 300
  * Purulent respiratory secretion)

SECONDARY OUTCOMES:
Duration of stay in ICU | up to 60 days
Duration of hospital say | up to 60 days
Sensitivity, specificity, and diagnostic accuracy of lung ultrasound to diagnose ventilator-associated pneumonia | up to 30 days
sensitivity, specificity, and diagnostic accuracy of lung ultrasound in association with the CPIS to diagnose ventilator-associated pneumonia | up to 30 days
sensitivity, specificity, and diagnostic accuracy of lung ultrasound in association with unprotected tracheal aspirate to diagnose ventilator-associated pneumonia | up to 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- GH Paris Saint Joseph, Paris, France
- Rianimazione I, (Dipartement of Anesthesia and Intensive Care Unit) of Fondazione IRCCS Policlinico S. Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bouhemad B, Liu ZH, Arbelot C, Zhang M, Ferarri F, Le-Guen M, Girard M, Lu Q, Rouby JJ. Ultrasound assessment of antibiotic-induced pulmonary reaeration in ventilator-associated pneumonia. Crit Care Med. 2010 Jan;38(1):84-92. doi: 10.1097/CCM.0b013e3181b08cdb. PMID 19633538
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Derived] Wang G, Ji X, Xu Y, Xiang X. Lung ultrasound: a promising tool to monitor ventilator-associated pneumonia in critically ill patients. Crit Care. 2016 Oct 27;20(1):320. doi: 10.1186/s13054-016-1487-y. PMID 27784331
- [Derived] Mongodi S, Via G, Girard M, Rouquette I, Misset B, Braschi A, Mojoli F, Bouhemad B. Lung Ultrasound for Early Diagnosis of Ventilator-Associated Pneumonia. Chest. 2016 Apr;149(4):969-80. doi: 10.1016/j.chest.2015.12.012. Epub 2015 Dec 22. PMID 26836896